CLINICAL TRIAL: NCT07150715
Title: Alpha-Emitting Radionuclide or Beta-Emitting Radionuclide Combined With Metastasis-Directed Stereotactic Body Radiotherapy for Oligorecurrent Prostate Adenocarcinoma (ANDROMEDA)
Brief Title: Alpha-Emitting Radionuclide or Beta-Emitting Radionuclide With Metastasis-Directed Stereotactic Body Radiotherapy for the Treatment of Recurrent, Oligometastatic Prostate Adenocarcinoma
Acronym: ANDROMEDA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-1338; NCI-2025-05583 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2025-08-25; First posted 2025-09-02 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Oligometastatic Prostate Adenocarcinoma; Recurrent Prostate Adenocarcinoma
MeSH Terms: interventions — (225)Ac-PSMA-617; Actinium; PSMA-617; Specimen Handling; gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11; Pluvicto; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm I (177Lu-PSMA-617) (Experimental): Patients receive 177Lu-PSMA-617 IV, over 1-10 minutes, on day one of each cycle. Cycles repeat every 6 weeks for 2 cycles. 4-6 weeks after completion of 177Lu-PSMA-617 patients receive 68Ga-PSMA-11 IV and undergo PSMA PET/CT scan. Within 4 weeks of the scan, patients receive SBRT, for 1-5 treatments, over 1- 1- days. Treatment is given in the absence of disease progression or unacceptable toxicity. Patients undergo PSMA PET/CT scan and blood sample collection throughout the study.
  Interventions: Drug: Actinium Ac 225 Vipivotide Tetraxetan; Procedure: Biospecimen Collection; Drug: Lutetium Lu 177 Vipivotide Tetraxetan; Procedure: PSMA PET-CT Scan; Radiation: Stereotactic Body Radiation Therapy
- Arm II (225Ac-PSMA-617) (Experimental): Patients receive 225Ac-PSMA-617 IV once. 4-6 weeks after completion of 225Ac-PSMA-617 patients receive 68Ga-PSMA-11 IV and undergo PSMA PET/CT scan. Within 4 weeks of the scan, patients receive SBRT, for 1-5 treatments, over 1- 1- days. Treatment is given in the absence of disease progression or unacceptable toxicity. Patients undergo PSMA PET/CT scan and blood sample collection throughout the study.
  Interventions: Drug: Actinium Ac 225 Vipivotide Tetraxetan; Procedure: Biospecimen Collection; Other: Gallium Ga 68 Gozetotide; Procedure: PSMA PET-CT Scan; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Actinium Ac 225 Vipivotide Tetraxetan — Given IV
  Other Names: 225Ac-labeled PSMA-617; 225Ac-PSMA-617; 225Ac-Vipivotide Tetraxetan; Actinium (225AC) PSMA-617; Actinium Ac 225 PSMA-617; Actinium Ac 225-PSMA-617; VIPIVOTIDE TETRAXETAN ACTINIUM AC-225
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Gallium Ga 68 Gozetotide — Given IV
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-DKFZ-PSMA-11; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA; 68Ga-PSMA-11; 68Ga-PSMA-HBED-CC; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; AAA 517; AAA-517; AAA517; Ga PSMA; Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled PSMA-11; GA-68 PSMA-11; Gallium Ga 68 PSMA-11; Gallium Ga 68-labeled PSMA-11; GALLIUM GA-68 GOZETOTIDE; Gallium-68 PSMA; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; GaPSMA; PSMA-HBED-CC GA-68
  Arms: Arm II (225Ac-PSMA-617)
Drug: Lutetium Lu 177 Vipivotide Tetraxetan — Given IV
  Other Names: 177Lu-labeled PSMA-617; 177Lu-PSMA-617; AAA 617; AAA-617; AAA617; Lu177-PSMA-617; Lutetium Lu 177-PSMA-617; LUTETIUM LU-177 VIPIVOTIDE TETRAXETAN; Lutetium-177-PSMA-617; Pluvicto
  Arms: Arm I (177Lu-PSMA-617)
Procedure: PSMA PET-CT Scan — Undergo PSMA PET/CT scan
  Other Names: PET-CT (PSMA); Prostate-specific Membrane Antigen PET-CT; PSMA PET-CT
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This phase II trial compares the use of 225Ac-PSMA-617 to 177Lu-PSMA-617, along with stereotactic body radiotherapy for the treatment of prostate cancer that has come back after a period of improvement (recurrent) and that has spread from where it first started (primary site) to multiple other places in the body (oligometastatic). 225Ac-PSMA-617 and 177Lu-PSMA-617 are radioactive drugs. They bind to a protein called a PSMA receptor, which is found on some prostate tumor cells. 225Ac-PSMA-617 or 177Lu-PSMA-617 builds up in these cells and gives off either alpha or beta radiation that may kill them. It is a type of radioconjugate and a type of PSMA analog. Stereotactic body radiation therapy (SBRT) is a type of external radiation therapy that uses special equipment to position a patient and precisely deliver radiation to tumors in the body (except the brain). The total dose of radiation is divided into smaller doses given over several days. This type of radiation therapy helps spare normal tissue. Giving 225Ac-PSMA-617 or 177Lu-PSMA-617 and metastasis directed stereotactic body radiotherapy may be effective in treating patients with recurrent, oligometastatic prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess progression-free survival for men with oligorecurrent prostate cancer after stereotactic body radiotherapy (SBRT) in combination with 2 cycles of Lutetium Lu 177 Vipivotide Tetraxetan (177Lu-PSMA-617) versus SBRT in combination with 1 cycle of Actinium Ac 225 Vipivotide Tetraxetan (225Ac-PSMA-617), with progression defined on the basis of prostate specific membrane antigen (PSMA) positron emission tomography (PET)/computed tomography (CT) scans obtained at 24 months post-SBRT or at the time of prostate specific antigen (PSA)-based biochemical progression, initiation of salvage therapy or death.

SECONDARY OBJECTIVES:

I. To evaluate burden of disease (including local control of irradiated lesions and presence of other disease) on a PSMA PET/CT obtained 24 months after SBRT + 177Lu-PSMA-617 versus SBRT + 225Ac-PSMA-617 in patients with oligometastatic disease who have not progressed by that point.

II. To assess physician-scored toxicity (common terminology criteria for adverse events [CTCAE] version 5.0) of SBRT + 177Lu-PSMA-617 versus SBRT + 225Ac-PSMA-617 in patients with oligometastatic disease.

III. To assess patient-reported quality of life (based on the Xerostomia Inventory scale) after SBRT + 177Lu-PSMA-617 versus SBRT + 225Ac-PSMA-617 in patients with oligometastatic disease.

IV. To assess androgen deprivation therapy (ADT)-free survival after 177Lu-PSMA-617 versus SBRT + 225Ac-PSMA-617 in patients with oligometastatic disease.

V. To determine local control of irradiated lesions at 24 months after last radionuclide infusion in patients with oligometastatic disease (based on a scheduled PSMA-PET), comparing 177Lu-PSMA-617 versus SBRT + 225Ac-PSMA-617.

VI. To assess time to locoregional progression, time to distant progression, time to new metastasis, and duration of response after last radionuclide infusion in patients with oligometastatic disease (as defined by PSMA PET/CT).

CORRELATIVE OBJECTIVES:

I. To quantitatively sequence T-cell receptor (TCR) repertoires using peripheral blood monocytes at baseline, 3 months, 6 months, and 12 months after last infusion of radionuclide.

II. To perform radiomics analysis on PSMA PET/CT scans performed at 24 months after last infusion of radionuclide, or at time of progression.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive 177Lu-PSMA-617 intravenously (IV) over 1-10 minutes on day one of each cycle. Cycles repeat every 6 weeks for 2 cycles. 4-6 weeks after completion of 177Lu-PSMA-617 patients receive Gallium Ga 68 Gozetotide (68Ga-PSMA-11) IV and undergo PSMA PET/CT scan. Within 4 weeks of the scan, patients receive SBRT for 1-5 treatments over 1- 1- days. Treatment is given in the absence of disease progression or unacceptable toxicity. Patients undergo PSMA PET/CT scan and blood sample collection throughout the study.

ARM II: Patients receive 225Ac-PSMA-617 IV once. 4-6 weeks after completion of 225Ac-PSMA-617 patients receive 68Ga-PSMA-11 IV and undergo PSMA PET/CT scan. Within 4 weeks of the scan, patients receive SBRT for 1-5 treatments, over 1- 1- days. Treatment is given in the absence of disease progression or unacceptable toxicity. Patients undergo PSMA PET/CT scan and blood sample collection throughout the study.

After completion of study treatment, patients are followed up every 3 months for 2 years and at 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Oligorecurrent prostate cancer as determined by the presence of 1-5 asymptomatic lesions outside the prostate or prostate bed identified on PSMA PET/CT by local readers
* Serum testosterone > 150 ng/dL
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* No indication for urgent or emergent radiation
* Histological confirmation of prostate adenocarcinoma (histology from original treatment acceptable)
* White blood cell count ≥ 2.5 × 109/L
* Platelets ≥ 100 × 109/L
* Hemoglobin ≥ 9 g/dL
* Total bilirubin ≤ 1.5 × institutional upper limits of normal (ULN) or up to 3 × ULN if known history of Gilbert's syndrome
* Alanine aminotransferase or aspartate aminotransferase ≤ 3.0 × ULN or ≤ 5.0 × ULN for patients with liver metastases
* Glomerular filtration rate creatinine-cystatin C (GFRcr-cys) ≥ 60 mL/min 1.73m2 using the Chronic Kidney Disease-Epidemiology Collaboration (CKD-EPI) 2021 equation
* Serum albumin > 3.0 g/dL
* Partner and patient must use a method of birth control with adequate barrier protection, deemed acceptable by the principal investigator during the study and for 3 months after last study drug administration
* Ability to understand, and willingness to sign, the written informed consent

Exclusion Criteria:

* Patients with neuroendocrine or small cell carcinoma of the prostate
* Patients with castrate-resistant disease (i.e., prostate specific antigen [PSA] > 0.5 ng/mL with serum testosterone <150 ng/dL)
* Patients who received androgen deprivation therapy or cytotoxic chemotherapy within 6 months of trial enrolment
* Concurrent systemic therapy for a solid organ malignancy
* Spinal cord compression
* Inability to lie flat
* Known hypersensitivity to components of 177-Lu-PSMA-617 or 225-Ac-Lu-PSMA-617
* Inadequate renal function of GFRcr-cys < 60 mL/min 1.73m2 using the CKD-EPI 2021equation
* Total bilirubin > 1.5 × ULN or > 3.0 × ULN if known history of Gilbert's syndrome
* Alanine aminotransferase or aspartate aminotransferase > 3 × ULN (or 5 × ULN for patients with known liver metastases)
* De novo oligometastatic disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2030-10-31 (Estimated); Study Completion 2031-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From the date of randomization to the date of disease progression or death, whichever happens earlier, up to 5 years
  A progression event will be based on prostate specific membrane antigen positron emission tomography/ computed tomography findings triggered either by a prostate specific antigen rise or at the timepoint defined by 24 months measured from the final radionuclide infusion (i.e., second infusion of 177Lu-PSMA-617 and first infusion of 225Ac-PSMA-617). The Kaplan-Meier (KM) method will be used to summarize PFS and log-rank test will be used to compare PFS between the two arms.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | From time of randomization, up to 5 years
  AEs will be summarized by type and grade.
Androgen deprivation therapy free survival | Up to 5 years
  The KM method will be used to summarize.
Time to locoregional progression | Up to 5 years
  The KM method will be used to summarize.
Time to new metastasis | Up to 5 years
  The KM method will be used to summarize.
Overall survival | Up to 5 years
  The KM method will be used to summarize.
Local control | Up to 5 years
  Will be defined based on PSMA PET/CT criteria, with scans obtained at time of PSA-progression of 24 months (if no progression by either time point). Patients with complete response, partial response, or stable disease will be considered as exhibiting local control. The proportion of lesions that have a stable or better response will be estimated using generalized estimating equation. The KM method will be used to summarize.
Duration of response over time | Up to 5 years
  The KM method will be used to summarize.
Quality of life as measured by xerostomia inventory | At baseline, 3 months, 6 months, 9 months, 12 months, 18 months, and 24 months
  Will be evaluated based on responses to the xerostomia inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Amar Kishan, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States